CLINICAL TRIAL: NCT00550654
Title: A Phase II Study of Hypofractionated Highly Conformal Radiation With Helical Tomotherapy for Extra-Cranial Oligo
Brief Title: Conformal Radiation Therapy in Treating Patients With Metastatic Cancer Outside the Brain
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was terminated due to poor accrual.
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Deborah Citrin, M.D., Principal Investigator, National Institutes of Health Clinical Center (CC)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 070230; NCI-07-C-0230
Record Dates: First submitted 2007-10-25; First posted 2007-10-30 (Estimated); Results first posted 2012-09-18 (Estimated); Last update posted 2017-01-13 (Estimated); Status verified 2016-11

CONDITIONS: Kidney Cancer; Melanoma (Skin); Metastatic Cancer; Ovarian Cancer; Sarcoma; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific; recurrent adult soft tissue sarcoma; recurrent melanoma; recurrent osteosarcoma; recurrent renal cell cancer; recurrent uterine sarcoma; stage IV adult soft tissue sarcoma; stage IV melanoma; stage IV uterine sarcoma; ovarian sarcoma; chondrosarcoma; metastatic osteosarcoma; stage IV renal cell cancer; lung metastases; liver metastases; bone metastases
MeSH Terms: conditions — Kidney Neoplasms; Melanoma; Neoplasm Metastasis; Ovarian Neoplasms; Sarcoma; Osteosarcoma; Carcinoma, Renal Cell; Chondrosarcoma | interventions — Radiotherapy, Conformal; Radiotherapy, Image-Guided; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Radiation Therapy in Metastatic Cancer (Experimental): Patients undergo hypofractionated highly conformal radiotherapy with helical tomotherapy once every other day over 5 days for a total of 3 fractions.
  Interventions: Other: questionnaire administration; Radiation: 3-dimensional conformal radiation therapy; Radiation: hypofractionated radiation therapy; Radiation: image-guided radiation therapy; Radiation: tomotherapy

INTERVENTIONS:
Other: questionnaire administration — Patients complete a pain assessment questionnaire, Brief Pain Inventory at baseline and at 1 and 3 months after treatment.
  Other Names: Brief Pain Inventory
Radiation: 3-dimensional conformal radiation therapy — Conformal radiation therapy improves the ability to spare normal tissues.
Radiation: hypofractionated radiation therapy — Hypofractionated radiation therapy is delivered to maximize pain relief while minimizing patient impact if life expectancy is short.
Radiation: image-guided radiation therapy — Image guided radiation therapy targets the specific site of disease.
Radiation: tomotherapy — Tomotherapy is a delivery method which provides megavoltage computed tomography (CT) localization and may provide superior conformality and localization compared to other dynamic intensity modulated radiation therapy techniques.

SUMMARY:
RATIONALE: Specialized radiation therapy that delivers a high dose of radiation directly to the tumor may kill more tumor cells and cause less damage to normal tissue.

PURPOSE: This phase II trial is studying how well conformal radiation therapy works in treating patients with metastatic cancer outside the brain.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To evaluate local control (defined as absence of local progression) at all treated sites of metastatic disease in patients with extracranial oligometastases treated with ablative doses of highly conformal radiotherapy delivered with helical tomotherapy.
* To evaluate local control at each treated site of metastatic disease in these patients.

Secondary

* To determine median time to local progression in patients treated with this regimen.
* To evaluate interfraction and intrafraction motion with megavoltage computed tomography (CT) imaging based on site of metastasis in these patients.
* To compare tumor growth during systemic therapy in tumors treated with targeted radiotherapy vs newly developed tumors that have not been treated with radiotherapy.
* To evaluate if treatment with hypofractionated highly conformal radiotherapy with helical tomotherapy can improve pain scores and decrease the need for analgesia in these patients.

OUTLINE: Patients are stratified according to histology (renal cell carcinoma vs melanoma vs sarcoma vs other histologies).

Patients undergo hypofractionated highly conformal radiotherapy with helical tomotherapy once every other day over 5 days for a total of 3 fractions. Patients undergo megavoltage imaging before and after each fraction to verify the positioning of each target lesion.

Patients complete a pain assessment questionnaire at baseline and at 1 and 3 months after treatment.

After completion of study therapy, patients are followed at 1 and 3 months and then every 3 months for up to 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Pathologically confirmed cancer

  * No active disease at the primary site as assessed by physical examination, clinical evaluation, or site-specific imaging
* Measurable metastatic disease meeting the following criteria:

  * Four or fewer sites of extracranial lesions < 5 cm in size
  * If metastatic site(s) is within the lung, the following criteria must be met:

    * No more than two metastases in the proximal bronchial tree area (defined as 2 cm from the trachea or mainstem bronchi)
    * Carbon monoxide diffusing capacity (DLCO) > 30% predicted and forced expiratory volume 1 (FEV1) > 1.2 L (in patients with more than one metastatic site in the lungs)
  * If metastatic site(s) is within 2 cm of either kidney, creatinine level must be < 1.5 times upper limit of normal (ULN)
  * If metastatic site(s) is within 2 cm of the liver, bilirubin level must be < 1.5 times ULN
* Patients with metastatic disease that meets any of the following criteria are excluded:

  * Proposed site(s) of treatment has been previously treated with radiotherapy
  * Metastatic site(s) requires emergent treatment (e.g., spinal cord compression, cauda equina, airway compromise, or life-threatening end-organ dysfunction)
  * Disease that is untreated or previously treated and progressive in the brain
  * Pathologic fracture or impending pathologic fracture at the metastatic site
  * Metastatic site(s) of a disease histology that is known to be sensitive to low doses of radiotherapy (e.g., pure seminoma, lymphoma, or small cell carcinoma)
* Patients in whom surgery is deemed an appropriate option as standard of care (e.g., isolated lung metastasis from sarcoma or isolated liver metastasis from colon cancer) but who refuse surgical therapy are eligible

PATIENT CHARACTERISTICS:

* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Life expectancy > 12 weeks as assessed by the consulting radiation oncologist
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No history of lupus erythematosus or scleroderma
* No known hypersensitivity to therapeutic radiotherapy
* No other malignancy within the past 2 years except nonmelanoma skin cancer or in situ malignancies of the cervix, bladder, or head and neck
* No unrelated systemic illness that, in the judgment of the investigator, would compromise the patient's ability to tolerate study therapy or would likely interfere with study procedures or results
* Able or likely to adhere to study treatment

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* More than 2 weeks since prior and no concurrent chemotherapy
* Prior or concurrent hormonal agents, including antiandrogens, gonadotropin-releasing hormone agonists, aromatase inhibitors, tamoxifen, or similar agents allowed
* No change in systemic therapy for 6 weeks before or within 4 weeks after initiating study radiotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2007-10; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deborah E. Citrin, MD, Principal Investigator — NCI - Radiation Oncology Branch; ROB
Locations (1):
- Warren Grant Magnuson Clinical Center - NCI Clinical Trials Referral Office, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Radiation Therapy in Metastatic Cancer
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Radiation Therapy in Metastatic Cancer
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.6 (NA) — It wasn't possible to calculate a standard deviation since there was only one participant.
Gender [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: 6-month Local Control (i.e., Complete Response, Partial Response, or Stable Disease) at All Treated Sites of Metastatic Disease
Description: Local control (e.g. absence of local progression) is defined as Complete response (CR), partial response (PR) or stable disease (SD) of the treated site(s). Complete response is the disappearance of the target lesion. Partial response is a >/= 50% decrease in maximal dimension compared to pretreatment imaging. Stable disease does not qualify for CR, PR, or progression.Progression is an interval increase in the maximal dimension of the target lesion.
Time Frame: 6 months
Population: No data/specimens were collected. Study was terminated due to poor accrual.
Arm/Group | Radiation Therapy in Metastatic Cancer
Number analyzed (Participants) | 0

2. Secondary Outcome: Number of Participants With Adverse Events
Description: Here is the number of participants with adverse events. For the detailed list of adverse events see the adverse event module.
Time Frame: 9 months, 11 days
Measure: Number; unit: Participants
Arm/Group | Radiation Therapy in Metastatic Cancer
Number analyzed (Participants) | 1
Participants | 1

3. Secondary Outcome: Median Time to Local Progression
Description: Interval from initiation of treatment on protocol to symptomatic or radiographic progression.
Time Frame: 6-12 months
Population: No data/specimens were collected. Study was terminated due to poor accrual.
Arm/Group | Radiation Therapy in Metastatic Cancer
Number analyzed (Participants) | 0

4. Secondary Outcome: 12 Month Local Control in All Sites of Treatment, and at Each Site of Treatment
Description: Local control (e.g. absence of local progression) is defined as Complete response (CR), partial response (PR) or stable disease (SD) of the treated site(s). Complete response is the disappearance of the target lesion. Partial response is a >/= 50% decrease in maximal dimension compared to pretreatment imaging. Stable disease does not qualify for CR, PR, or progression. Progression is an interval increase in the maximal dimension of the target lesion.
Time Frame: 12 months
Population: No data/specimens were collected. Study was terminated due to poor accrual.
Arm/Group | Radiation Therapy in Metastatic Cancer
Number analyzed (Participants) | 0

5. Secondary Outcome: Interfraction and Intrafraction Motion With Megavoltage Computed Tomography (CT) Based on Sites of Metastasis
Description: Megavoltage localization scans will be obtained and the physician and therapist will evaluate the cone beam image and compare this image to the expected image based on the patient's initial planning CT scan.
Time Frame: One to three months of followup
Population: No data/specimens were collected. Study was terminated due to poor accrual.
Arm/Group | Radiation Therapy in Metastatic Cancer
Number analyzed (Participants) | 0

6. Secondary Outcome: Pain at Sites of Metastases
Description: Improvement in pain from baseline will be assessed by the Brief Inventory for Pain criteria.
Time Frame: One and three months of follow up
Population: No data/specimens were collected. Study was terminated due to poor accrual.
Arm/Group | Radiation Therapy in Metastatic Cancer
Number analyzed (Participants) | 0

7. Secondary Outcome: Tumor Doubling Times During Systemic Treatment Compared Between Tumors Untreated With Radiation (Newly Developed Tumors) and Tumors Which Have Received Radiation Therapy
Description: Rate of growth of the composite (total) treated volume (up to four sites) compared to the composite volume of up to four newly identified and untreated prospectively-identified (at the time of systemic progression) metastatic sites. Volume doubling time will be calculated assuming an exponential growth pattern.
Time Frame: Baseline and prior to termination of systemic therapy or protocol withdrawal
Population: No data/specimens were collected. Study was terminated due to poor accrual.
Arm/Group | Radiation Therapy in Metastatic Cancer
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Radiation Therapy in Metastatic Cancer
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Radiation Therapy in Metastatic Cancer (N=1)
Pain::Buttock (Musculoskeletal and connective tissue disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Urinary retention (including neurogenic bladder) (Renal and urinary disorders) | 1 (1)
Weight loss (General disorders) | 1 (1)
Dermatology/Skin - Other (Specify) (Skin and subcutaneous tissue disorders) | 1 (1)
Anorexia (Gastrointestinal disorders) | 1 (1)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 1 (1)
Taste alteration (dysgeusia) (Gastrointestinal disorders) | 1 (1)
Pain::Extremity-limb (Musculoskeletal and connective tissue disorders) | 1 (1)
Hemorrhage, pulmonary/upper respiratory: Nose (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No